CLINICAL TRIAL: NCT07018232
Title: Enhancing Timely Access to Medication Changes: The Role of Ambulatory Care Pharmacists in Overcoming Transitions of Care Challenges
Brief Title: Enhancing Timely Access to Medication Changes: The Role of Pharmacists in Overcoming Transitions of Care Challenges
Status: Completed | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2411-102
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Transitional Care
Keywords: pharmacist; medication access; hospital discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medication Gap: A patient with a medication gap was defined as 1) having lapse in prescription coverage or any number of days where they were out of a maintenance prescription medication because the primary care provider did not send in a refill in time, and 2) having a medication access barrier, such as needing to contact the primary care provider to send in a refill for a maintenance prescription medication.
  Interventions: Behavioral: Unplanned healthcare encounter
- No Medication Gap: A patient with no medication gap was defined as having zero days without a maintenance prescription medication because it was appropriately refilled by their primary care provider at a transitions of care follow-up appointment
  Interventions: Behavioral: Unplanned healthcare encounter

INTERVENTIONS:
Behavioral: Unplanned healthcare encounter — Patient needing to connect with healthcare to fill a medication gap

SUMMARY:
Objective: Among patients discharged from the hospital with changes in maintenance prescription medication, how does experiencing a medication access gap compared to a no medication access gap impact the time to first unplanned healthcare encounter?

This is a retrospective, cohort study conducted at two hospital sites in rural Pennsylvania and New York State using encounter data from the electronic health record to analyze any patient discharged with medication changes from June 1, 2023 to May 31, 2024.

DETAILED DESCRIPTION:
Background: Transitions of care are high-risk periods marked by frequent medication-related problems with up to 80% of discharged patients and 98% of older adults experiencing discrepancies in their medication regimens. These gaps, often due to delayed prescription refills or poor care coordination, contribute to unplanned healthcare encounters, increased costs, and strain on providers. Pharmacists can mitigate these risks by improving medication access and continuity.

Objective: Among patients discharged from the hospital with changes in maintenance prescription medication, how does experiencing a medication access gap compared to a no medication access gap impact the time to first unplanned healthcare encounter?

This is a retrospective, cohort study conducted at two hospital sites in rural Pennsylvania and New York State using encounter data from the electronic health record to analyze any patient discharged with medication changes from June 1, 2023 to May 31, 2024.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Have a Guthrie primary care provider
* Discharged from the hospital to home or self-care (routine)
* Had a medication change on discharge based on a discharge summary and/or after visit summary (AVS) containing "start taking these medications", "continue these medications which have changed", and/or "stop taking these previous medications".

Exclusion Criteria:

* Age less than 18 years of age
* Do not have a Guthrie primary care provider
* Discharged from the hospital to anywhere besides home or self-care (routine) such as to rehabilitation, long-term care, left against medical advice, or transferred to another type of healthcare institution
* prescriptions on discharge that lack e-prescribing class
* prescriptions on discharge for day supplies less than 28 days
* prescriptions on discharge for day supplies greater than 45 days
* prescriptions on discharge with 1 or more refills provided
* prescriptions on discharge for as needed medications
* prescriptions on discharge for anti-infective agent
* prescriptions on discharge for short-term steroids
* prescriptions on discharge for nausea medication
* prescriptions on discharge for bowel regimen medication
* prescriptions on discharge for diabetic or medical supplies
* prescriptions on discharge for topical medications
* prescriptions on discharge for cough suppressants,
* prescriptions on discharge for vitamins and supplements
* prescriptions on discharge for medications that can be purchased over the counter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients discharged from an acute care hospital with a change in their chronic prescription medication regimen
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Number of days to first unplanned healthcare encounter post-discharge | 90 days after discharge
  The study will compare number of days between patients who had a medication gap and patients who had no medication gap

SECONDARY OUTCOMES:
Number of days that a patient is without a prescribed medication post-discharge | 90 days after discharge
  The study will compare the number of days patients are without a prescribed medication after hospital discharge, for the two groups (1 patients who had a medication gap and 2 patients who had no medication gap).
Describe the types of drug-related problems and/or medication access barriers between the two groups | 90 days after discharge
  The study will compare the types of drug-related problems and medication access barriers between the two groups (1 patients who had a medication gap and 2 patients who had no medication gap).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Van Dyke, PharmD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No